CLINICAL TRIAL: NCT06826209
Title: Comparison of Upper Extremity Functional Performance, Muscle Strength, and Activities of Daily Living Levels in Children with Hemophilia and Healthy Children
Brief Title: Comparison of Upper Extremity Functional Performance in Hemophilic and Healthy Children
Status: Enrolling by invitation | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ferhat Öztürk, Researcher, Hacettepe University
Other Study IDs: FTREK24/103
Record Dates: First submitted 2025-02-06; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Hemophilia; Upper Extremity; Strength; Performance; Children
Keywords: Hemophilia; Muscle Strength; Upper Extremity
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hemophilia groups: Patients group

SUMMARY:
The goal of this observational study is to evaluate the functional performance of the upper extremity joints (scapula, shoulder, elbow, and wrist) in haemophilic children and compare muscle strength and ADL limitations with healthy children.

DETAILED DESCRIPTION:
This study aims to evaluate the upper extremity functional performance, muscle strength, and daily living activity levels of hemophilic children and compare them with healthy children. The goal is to determine the effects of hemophilia on these children and contribute to the development of appropriate rehabilitation strategies. Parameters include explosive strength, isometric muscle strength, wrist grip strength, and functional exercise capacity. Additionally, the ADL-Glittre pediatric version test and Hemophilia Joint Health Score (HJHS) will be used to assess joint health and GYA performance. Muscle strength is crucial for hemophilic children to perform daily activities, and the relationship between muscle strength and GYA levels will be investigated. The project aims to guide the development of physiotherapy and rehabilitation strategies for hemophilic children and contribute to the literature by filling existing gaps, ultimately creating an important reference for healthcare professionals and families.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Hemophilia A or B
* Receiving prophylaxis treatment (a routine treatment)
* Negative for inhibitors at the time of enrollment

Exclusion Criteria:

* Positive for inhibitors at the time of enrollment
* Acute elbow bleeding
* History of acute muscle bleeding
* History of surgery in any upper extremity joints
* Having undergone radionuclide synovectomy

Ages: 7 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Male children diagnosed with Hemophilia, who are being followed by the same physician at the Hematology Unit of the Department of Pediatrics, Faculty of Medicine, Hacettepe University, will be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2026-06-24 (Estimated); Study Completion 2026-10-24 (Estimated)

PRIMARY OUTCOMES:
Hemophilia Joint Health Score | Through study completion, an average of 1 year
  The Hemophilia Joint Health Score (HJHS) is a clinical tool used to assess joint health in individuals with hemophilia, focusing on major joints such as the knees, elbows, and ankles. It evaluates symptoms like pain, swelling, and range of motion restrictions, with a grading system that helps determine the severity of joint damage. The HJHS also considers joint function in daily activities, making it an essential tool for monitoring joint health and the progression of hemophilic arthropathy. It plays a vital role in both clinical management and research, helping guide treatment strategies and assess their effectiveness.

SECONDARY OUTCOMES:
Muscle Strength | Through study completion, an average of 1 year
  The Lafayette Handheld Dynamometer is a device used to measure upper extremity muscle strength in children with hemophilia. It assesses muscle strength under isometric conditions and is typically used to test the muscles around the shoulder, elbow, and wrist. The measurements aim to determine the maximum force exerted by the muscles, which is important for identifying potential reductions in muscle strength in individuals with hemophilia. This test is valuable for determining physical performance levels, planning treatment approaches, and guiding rehabilitation processes.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe Universit, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Undecided